CLINICAL TRIAL: NCT00695149
Title: Clinical Study of Treatment for Acute Spinal Cord Injury Using Cultured Bone Marrow Stromal Cells
Brief Title: Treatment for Acute Spinal Cord Injury
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHA_SCI0401
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord Injury; Central nervous system; Regeneration; Bone marrow stromal cells; Transplantation
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Transplantation of bone marrow stromal cell

SUMMARY:
This clinical trial aims to treat a damaged spinal cord by injecting your own bone marrow stromal cells (autologous bone marrow stromal cells) into cerebrospinal fluid through the lumbar puncture, and assess the safety and efficacy of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury is confirmed with MRI
* Methylprednisolone therapy according to this study can be started within 8 hours after the injury
* Bone marrow stromal cells (BMSCs) incubation can be started within 72 hours after the injury
* Age between 15 and 60
* With the informed consent of obtaining bone marrow and injecting incubated BMSCs.

Exclusion Criteria:

* Complete disruption of spinal cord
* Central spinal cord injury
* Spinal canal stenosis before the injury
* Brain or spinal cord disease before the injury
* Positive serologic test in at least one of the following; HBs antigen, HCV antibody, HIV antibody, or HTLV-1 antibody
* Pregnancy

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Motor function | six months

SECONDARY OUTCOMES:
Sensation | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Kansai Medical University, Moriguchi, Osaka, Japan

REFERENCES:
- [Background] Ohta M, Suzuki Y, Noda T, Ejiri Y, Dezawa M, Kataoka K, Chou H, Ishikawa N, Matsumoto N, Iwashita Y, Mizuta E, Kuno S, Ide C. Bone marrow stromal cells infused into the cerebrospinal fluid promote functional recovery of the injured rat spinal cord with reduced cavity formation. Exp Neurol. 2004 Jun;187(2):266-78. doi: 10.1016/j.expneurol.2004.01.021. PMID 15144853
- [Derived] Saito F, Nakatani T, Iwase M, Maeda Y, Murao Y, Suzuki Y, Fukushima M, Ide C. Administration of cultured autologous bone marrow stromal cells into cerebrospinal fluid in spinal injury patients: a pilot study. Restor Neurol Neurosci. 2012;30(2):127-36. doi: 10.3233/RNN-2011-0629. PMID 22232031